CLINICAL TRIAL: NCT06155383
Title: A Phase II Study of Perioperative Disitamab Vedotin Plus Toripalimab and XELOX Versus Disitamab Vedotin Plus Toripalimab Versus XELOX in Subjects With HER2-expressing Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma.
Brief Title: Perioperative Disitamab Vedotin Plus Toripalimab and XELOX in Gastric or Gastroesophageal Junction Adenocarcinoma.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C022
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: HER2-expressing; gastric cancer; gastroesophageal junction adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin; disitamab vedotin; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- XELOX (capecitabine + oxaliplatin) (Active Comparator): capecitabine with oxaliplatin arm
  Interventions: Drug: Capecitabine; Drug: oxaliplatin
- Disitamab Vedotin + Toripalimab (Experimental): Disitamab Vedotin with Toripalimab arm
  Interventions: Drug: Disitamab Vedotin; Drug: Toripalimab
- Disitamab Vedotin + Toripalimab + XELOX (Experimental): Disitamab Vedotin + Toripalimab + XELOX arm
  Interventions: Drug: Capecitabine; Drug: oxaliplatin; Drug: Disitamab Vedotin; Drug: Toripalimab

INTERVENTIONS:
Drug: Capecitabine — 1000 mg/m2, Bid orally, D1-14, every 3 weeks
  Arms: Disitamab Vedotin + Toripalimab + XELOX; XELOX (capecitabine + oxaliplatin)
Drug: oxaliplatin — 130 mg/m2, intravenous infusion, D1, every 3 weeks
  Arms: Disitamab Vedotin + Toripalimab + XELOX; XELOX (capecitabine + oxaliplatin)
Drug: Disitamab Vedotin — 2.5 mg/kg, intravenous infusion, D1, every 2 weeks
  Other Names: RC48
  Arms: Disitamab Vedotin + Toripalimab; Disitamab Vedotin + Toripalimab + XELOX
Drug: Toripalimab — 3.0 mg/kg, intravenous infusion, D1, every 2 weeks
  Other Names: JS001
  Arms: Disitamab Vedotin + Toripalimab; Disitamab Vedotin + Toripalimab + XELOX

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of perioperative Disitamab Vedotin plus Toripalimab and XELOX versus Disitamab Vedotin plus Toripalimab versus XELOX in subjects with HER2-expressing resectable locally advanced gastric or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
This is an open-label, randomized, multicenter, open-label clinical trial designed to evaluate safety and efficacy of perioperative Disitamab Vedotin plus Toripalimab and XELOX versus Disitamab Vedotin plus Toripalimab versus XELOX in subjects with HER2-expressing (immunohistochemical 1+, 2+, 3+) resectable locally advanced gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign the informed consent form;
2. Male or female, ≥18 years;
3. Patients with gastric or gastroesophageal junction adenocarcinoma confirmed by histopathology;
4. Clinical stage cT3-4aN+, no distant metastasis (M0);
5. According to the baseline imaging and medical history data evaluated by the Investigators, radical surgery for gastric cancer and R0 resection is expected; Subjects had not previously received any antitumor therapy for gastric or gastroesophageal junction adenocarcinoma;
6. HER2- expression: IHC 1+, 2+, 3+;
7. ECOG performance status score of 0 or 1;
8. Cardiac function: left ventricular ejection fraction ≥50%;
9. The following criteria should be met within 7 days prior to study dosing (normal values are based on the clinical trial center):

   9.1Bone marrow function:
   1. absolute neutrophil count (ANC) ≥1.5×109/L (no treatment with granulocyte colony-stimulating factor within 1 week prior to examination);
   2. Platelets ≥100×109/L (platelets should not be transfused within 1 week before the examination, and recombinant human thrombopoietin therapy should not be used within 2 weeks)
   3. hemoglobin ≥9g/dL (blood transfusion and erythropoietin treatment are not allowed within 2 weeks prior to the examination);

   9.2Liver function:
   1. Serum total bilirubin ≤1.5 times the upper limit of normal (ULN);
   2. alanine amino transferase (ALT) and aspartate amino transferase (AST) ≤2.5 × ULN;

   9.3 Kidney function:

   a.Blood creatinine ≤1.5×ULN or creatinine clearance (CrCl) ≥50 mL/min according to Cockcroft-Gault formula method; Female: CrCl= (140-age) × weight (kg) × 0.85 72 × serum creatinine (mg/dL) Male: CrCl= (140-age) × weight (kg) × 1.00 72 × serum creatinine (mg/dL)

   9.4 Coagulation function:
   1. prothrombin time (PT) ≤1.5×ULN;
   2. thrombin time (TT) ≤ 1.5×ULN;
   3. activated partial thromboplastin time (APTT) ≤ 1.5×ULN.
10. Female subjects should be surgically sterilized, postmenopausal, or agree to use at least one medically acceptable method of contraception (e.g., intrauterine device, contraceptives, or condoms) for 7 days before the first dose and for 6 months after the end of the study treatment period, and not breastfeed. Blood pregnancy tests must be negative within 7 days prior to study enrollment. Male subjects should agree to use at least one medically approved contraceptive method (e.g., condoms, abstinence, etc.) for 7 days prior to initial dosing and up to 6 months after the end of the study treatment period;
11. Able to understand trial requirements, willing and able to follow trial and follow-up procedures.

Exclusion Criteria:

1. Received any anti-tumor therapy for gastric or gastroesophageal junction adenocarcinoma before study dosing, including chemotherapy, radiotherapy, targeted therapy, immunotherapy and other anti-tumor drug therapy (including Chinese medicine treatment with anti-tumor ingredients specified in the instructions within 2 weeks before screening);
2. The investigators considered perioperative period treatment of patients requiring radiotherapy for target lesions；
3. Major surgery was performed within 4 weeks before the start of study dosing and did not fully recover;
4. Patients with active gastrointestinal bleeding or high risk of bleeding within 2 weeks prior to screening;
5. Gastrointestinal perforation/fistula 6 months before screening;
6. Upper digestive tract obstruction that cannot guarantee drug absorption, functional abnormalities or malabsorption syndrome, which can affect the absorption of capecitabine ;
7. Peripheral polyneuropathy ≥ NCI Ⅱ grade；
8. Serum virology examination (based on the normal value of the research center):

   * Positive HBsAg test with positive HBV DNA copy number;
   * Positive HCVAb test with positive HCV RNA PCR test.
   * Positive HIVAb test.
9. Have received live vaccine within 4 weeks prior to screening or plan to receive any vaccine during the study period (except for the novel coronavirus vaccine);
10. Heart failure rated 3 or higher by the New York College of Cardiology (NYHA);
11. Cardiac chest pain, defined as moderate pain that restricts daily activities, occurred within 28 days prior to screening. There were serious arteriovenous thrombosis events or cardiovascular and cerebrovascular accidents within six months before dosing, such as deep vein thrombosis (except asymptomatic and untreated intermuscular venous thrombosis), pulmonary embolism, cerebral infarction, cerebral hemorrhage, and myocardial infarction (except asymptomatic lacunar infarction that did not require clinical intervention);
12. There is an active or advanced infection that requires systematic treatment (experimental medication may be initiated 2 weeks after the end of anti-infective therapy), such as active tuberculosis;
13. There are systemic diseases that have not been stably controlled which are determined by investigators, including diabetes, hypertension, cirrhosis, etc.;
14. A history of lung disease that requires treatment and has the potential to interfere with surgery, including but not limited to interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis, and acute lung disease;
15. Active autoimmune diseases requiring systemic therapy (such as the use of disease-modifying drugs, corticosteroids, or immunosuppressive drugs) within 2 years prior to dose administration, and replacement therapies (e.g., thyroxine, insulin, or physiological replacement of glucocorticoids due to renal or pituitary deficiency) are allowed, and a history of refractory autoimmune disease. Systemic use of steroids within 14 days prior to screening (dose > 10 mg/day prednisone or equivalent dose of other glucocorticoids) or other systemic immunosuppressive therapy;
16. Other malignancies within 5 years prior to screening, other than those that have been cured after treatment (including but not limited to adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or breast ductal carcinoma in situ treated with radical surgery);
17. Previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
18. Allergies to any of the drugs in this study;
19. Known deficiency of dipyrimidine dehydrogenase (DPD);
20. Receiving immunotherapy (including but not limited to interleukin, interferon, thymus hormone) or other investigational drugs within 28 days prior to screening;
21. Pregnant or lactating women;
22. Any other disease, metabolic disorder, or abnormal findings upon physical examination or laboratory examination that makes the subject unsuitable for receiving the investigational drug, affects the interpretation of study outcomes, or poses risks to patient safety, as determined by the investigator;
23. Subject is assessed to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Up to approximately 2 years
  Proportion of patients with pCR. pCR is defined as no invasive disease within an entirely submitted and evaluated gross lesion, and histologically negative nodes (ypT0N0)

SECONDARY OUTCOMES:
Objective remission rate (ORR) | Up to approximately 2 years
  The objective response rate will be mainly analyzed by according to the RECIST 1.1 standard tumor evaluation by the investigator will be performed).
R0 resection rate | Up to approximately 2 years
  Percentage of patients with complete resection of tumor tissue without tumor cell infiltration at surgical margins
Tumor regression grade (TRG) score | Up to approximately 2 years
  to evaluate tumor regression grade (based on postoperative pathological reports);
Major pathological response (MPR) | Up to approximately 2 years
  the proportion of patients with percentage of residual tumor cells in the tumor bed ≤10% after neoadjuvant therapy;
Event free survival (EFS) | Up to approximately 2 years
  the time from randomization to the first occurrence of the following events: radiographic disease progression per RECIST 1.1,local or distant recurrence, and death due to any cause;
Overall survival (OS) | Up to approximately 2 years
  OS is defined as the time from randomization to death due to any cause.
Adverse events | Time Frame: Up to approximately 2 years
  to evaluate safety including adverse event rate and adverse event grade

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Fang, Ph.D, Study Director — RemeGen Co., Ltd.
Locations (11):
- China (11):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Yunnan Cancer Hospital, Kunming, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Shandong Cancer Hospital & Institute, Jinan, Shangdong
  - Sichuan Cancer Hospital & Institute, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No